CLINICAL TRIAL: NCT06964581
Title: Cognitive Rehabilitation of Deficits in Patients With Multiple Sclerosis: Proposal for an Integrated Cognitive Treatment in a Telematic Format
Brief Title: Cognitive Rehabilitation of Deficits in Patients With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Valentina Varalta, Doctor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3995CESC
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Telerehabilitation; Multiple Sclerosis; Cognitive Disorders; Neurorehabilitation
Keywords: telerehabilitation; multiple sclerosis; cognitive disorders
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Three hours of cognitive rehabilitation per week, carried out independently and remotely using a computerized device, which is pre-programmed according to the patient's specific needs.
  Interventions: Behavioral: Cognitive treatment delivered via telerehabilitation.
- In-person treatment (Active Comparator): Three hours of in-person cognitive rehabilitation per week using a computerized device. The participant will perform cognitive exercises on the computerized device in the presence of the therapist, who will activate the device (using credentials specifically created for them) and select the appropriate activity to administer at each session.
  Interventions: Behavioral: In-person cognitive treatment.

INTERVENTIONS:
Behavioral: Cognitive treatment delivered via telerehabilitation. — Three hours of cognitive rehabilitation per week, carried out independently and remotely using a computerized device, which is pre-programmed according to the patient's specific needs.
  Arms: Telerehabilitation
Behavioral: In-person cognitive treatment. — Three hours of in-person cognitive rehabilitation per week using a computerized device. The participant will perform cognitive exercises on the computerized device in the presence of the therapist, who will activate the device (using credentials specifically created for them) and select the appropriate activity to administer at each session.
  Arms: In-person treatment

SUMMARY:
Non-Inferiority Study, Post-Market Clinical Investigation with a Device, Single-Blind Randomized Controlled Trial in a Cohort of Patients Diagnosed with Multiple Sclerosis (MS).

The aim of the study is to assess whether a computer-based cognitive treatment delivered via telerehabilitation produces effects from T0 to T1 that are not inferior to those of an in-person treatment on sustained attention in a cohort of patients with MS.

The secondary objective is to evaluate the effects of telerehabilitation compared to the same treatment delivered in person on attentional shifting, memory, executive functions, and daily functioning (including cognitive fatigue, quality of life, and mood) in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting multiple sclerosis (RRMS), or primary progressive (PPMS) or secondary progressive (SPMS), defined by at least 3-6 months.
* Age between 18 and 65 years.
* Expanded Disability Status Scale (EDSS) between 3 and 5 to include patients with overall neurological disability from mild to moderate.
* Presence of one or more of the following cognitive disorders (reported by the patient and subsequently confirmed through the Oxford Cognitive Screen-OCS):
* Memory disorders
* Attention disorders
* Executive function disorders
* Availability of internet at the patient's home necessary for the tele-rehabilitation procedures.
* Adequate visual and auditory abilities to use the rehabilitation device.

Exclusion Criteria:

* Presence of other neurological conditions;
* Psychiatric disorders in medical history;
* Alcohol and/or drug abuse;
* Presence of uncorrected severe visual deficits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Paced Auditory Serial Addition Task (PASAT) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  In the Paced Auditory Serial Addition Task (PASAT), the patient listens to a recorded voice reading a series of numbers at regular intervals. They must mentally add each number to the one immediately preceding it and respond orally. The test assesses sustained attention, working memory, and processing speed. The maximum score, usually 60, corresponds to the number of correct responses, with higher scores indicating better cognitive performance.

SECONDARY OUTCOMES:
Trail Making Test Part A (TMT-A) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Trail Making Test Part A (TMT-A) is a neuropsychological assessment that measures selective attention and processing speed. Participants connect a series of numbered circles in sequential order as quickly as possible. The score is determined by the time taken to complete the task, with shorter times indicating better performance. Errors may negatively impact the score.
Trail Making Test Part B (TMT-B) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Trail Making Test Part B (TMT-B) is a neuropsychological test that measures Divided attention. Participants must connect numbered and lettered circles in alternating order as quickly as possible. The score is based on the time taken to complete the test, with shorter times indicating better performance. Any errors may negatively impact the score.
Symbol Digit Modalities Test | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  This test evaluates the visual information processing speed and attention; the number of correct answers in 90 seconds is registered (higher scores indicate better performance).
Modified Five Point Test (MFPT) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Modified Five Point Test (MFPT), which is a measure of figural fluency assessing the ability to initiate mental productivity and self-monitoring during a visual-spatial task. Performance is assessed by scoring the total number of correct and unique designs generated in 3 min (UDs), and the total number of UDs produced into strategies (CSs).
"Learning" subtest of the Rivermead Behavioural Memory Test-3 (RBMT-3) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  "Learning" subtest of the Rivermead Behavioural Memory Test-3 (RBMT-3), used to assess the ability to learn and recall visuospatial information after a delay. The learning trial has a score range of 0 to 51 correct items, and the delayed recall trial ranges from 0 to 17 correct items, with higher scores indicating better performance.
Phonemic Verbal Fluency Test | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Phonemic Verbal Fluency Test is used to investigate the ability to access the semantic-lexical store (number of items, with higher scores indicating better performance).
Test of Attentional Performance (TAP) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Test of Attentional Performance (TAP) is used to assess reaction times ("Alertness") and the ability to inhibit automatic responses ("Go/No-Go") (reaction times, with higher scores indicating worse performance).
Modified Fatigue Impact Scale (MFIS) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Modified Fatigue Impact Scale (MFIS) is used to evaluate the degree of fatigue (range 0-84, with higher scores indicating worse performance).
Multiple Sclerosis Quality of Life 54 (MSQOL-54) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Multiple Sclerosis Quality of Life 54 (MSQOL-54) is used to assess quality of life (range varies by item, with higher scores indicating better performance).
Depression, Anxiety, and Stress Scale (DASS) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Depression, Anxiety, and Stress Scale (DASS) is used to evaluate psychological well-being (range 0-63, with higher scores indicating worse performance).

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona - UOC di Neuroriabilitazione, Verona, verona, Italy